CLINICAL TRIAL: NCT06343610
Title: The Effect of 8-week Dietary Intake of Novel Food Supplement on Minimal Erythema Dose: Randomised Double Blind, Placebo-controlled Study
Brief Title: The Effect of 8-week Dietary Intake of Novel Food Supplement on Minimal Erythema Dose
Acronym: VIST-TO-UV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIST TO-UV 01-2024
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Minimal Erythema Dose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator)
  Interventions: Dietary Supplement: Active product
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active product — Contains a complex of: Calaguala leaves extract (Polypodium leucotomos), vitamin C (L-ascorbic acid), blood orange fruit extract (Citrus sinensis; red orange extract), vitamin E (alpha-tocopheryl acetate), vitamin A (retinyl palmitate), vitamin D3 cholecalciferol.
  Arms: Test group
Dietary Supplement: Placebo — No active ingredients.
  Arms: Placebo group

SUMMARY:
This is a double-blind, randomized, placebo-controlled interventional study of the effect of multiple-dose dietary intake on minimal erythema dose and other skin parameters.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled interventional study of the effect of multiple-dose dietary intake on minimal erythema dose and other skin parameters.

The study will be performed on 54 adults, between the ages 21 and 65 years and will include daily dietary supplementation over 8-weeks period.

Participants will be randomly assigned in one of two groups, 27 in each. One group (test group) will receive investigational product, a syrup containing red orange extract, Calaguala extract and vitamins A, C, D, E and the other placebo syrup. Participants will continuously receive placebo or investigational product for 8 weeks in order to determine multiple-dose effects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian volunteers aged between 21 and 65 years at the time of the signature of Informed consent form (ICF),
* Signed Informed consent form (ICF),
* Fitzpatrick skin phototypes I-III,
* No skin pigmentation disorders,
* In good health condition,
* Willingness to avoid a consumption of any food supplements containing red orange extract, polypodium extract, carotenes or other antioxidants that could interfere with the results during the study,
* Willingness to avoid the sun, tanning beds and tanning products on the test area during the study,
* Willingness to follow all study procedures and keeping a diary during the study (to follow their compliance and palatability),
* No changes in dietary habits or dietary supplements in last 2 months prior to inclusion.
* No changes in cosmetic body care routine in last month prior to inclusion on measurement areas.
* No recent participation in any other similar study.
* No sun exposure (both natural and artificial) for at least two months before study start on the test area.
* Absence of sunburn, suntan, scars, or other active dermal lesions on the test area.
* Colour uniformity of the test area (without tattoo, nevi, blemishes or solar lentigo and without hair).

Exclusion Criteria:

* Pregnancy or breastfeeding or planning pregnancy in next 6 months (for women)
* Known or suspected allergy to any ingredient of the tested products or UV radiation.
* Dermatological problems in the test area or the requirement for annual mole checks by a dermatologist.
* Pharmacological treatments (both locally or systemically) that could interfere with the results.
* Positive anamnesis for atopy (allergic hypersensitivity affecting parts of the body not in direct contact with the allergen)
* Use of self-tanning products for at least 2 months before study start.
* Medication with photosensitizing potential, drugs, corticoids in last month prior to study start.
* Regular consumption of food supplements containing red orange extract, polypodium extract, carotenoids or other antioxidants or supplements able to induce skin colour in last month before inclusion into the study.
* Any clinically significant history of melanoma or skin cancer (including their immediate family), serious metabolic disease, digestive tract disease, liver disease, kidney disease, haematological disease or other illness that could interfere with the study.
* History of severe reactions from exposure to sunlight (i.e., polymorphous light eruption)
* Any surgery, chemical or physical treatment on the experimental area within the 12 months prior to the study or foreseeing it for the duration of the study.
* Regular depilation of test area.
* Planning a hospitalization during the study.
* Impaired immune system due to autoimmune diseases, or use of immunosuppressive medication.
* Mental incapacity that precludes adequate understanding or cooperation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change of minimal erythema dose | 8 weeks
  Increase of minimal erythema dose (MED) from baseline in test group in comparison to placebo group. Irradiation for determination of MED (J/cm2), will be performed with automated erythema tester Dermalight® 80 MED Tester (Dr Hoenle Medizintechnik GmbH, Germany; UVB 311 nm).

SECONDARY OUTCOMES:
Change of redness formation | 8 weeks
  Decrease of redness formation following UVB irradiation in test group in comparison to placebo group. Redness measurements (CIE a*) will be done before irradiation and after 24 hours post irradiation and variation of a* calculated for each of the follow-up visits before and after 8 weeks of supplementation. The skin colour will be measured by Cortex Colorimeter DSM-4 (Cortex Technology ApS, Denmark). The colorimeter uses CIE L* a* b* tridimensional colour space; a* values (red-green axis) are an indicator of erythema/redness formation.

OTHER OUTCOMES:
Change of melanin index | 8 weeks
  Change of melanin index (MI) following UVB irradiation in test group in comparison to placebo group. MI measurements will be done before irradiation and after 48 hours post irradiation and variation of MI calculated for each of the follow-up visits before and after 8 weeks of supplementation. MI will be measured by Cortex Colorimeter DSM-4 (Cortex Technology ApS, Denmark). The colorimeter uses CIE L* a* b* tridimensional colour space. MI is a measure of pigmentation of the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- VIST - Faculty of Applied Sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No